CLINICAL TRIAL: NCT03715647
Title: Correlation of the Driving Pressure With the Survival of Puerperae Under Mechanical Ventilation by Electrical Impedance Tomography
Brief Title: Correlation of Survival in Puerperae by Electrical Impedance Tomography
Acronym: COSIPBEIT
Status: Completed | Type: Observational
Sponsor: Amazon University (Other)
Collaborators: Santa Casa de Misericórdia do Pará (Unknown)
Responsible Party: Principal Investigator, Paulo Eduardo Santos Avila, Assistant teacher, Amazon University
Other Study IDs: 2.251.640
Record Dates: First submitted 2018-07-25; First posted 2018-10-23 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Postpartum Period; Sepsis; Respiratory Distress Syndrome,Adult; HELLP Syndrome
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome; HELLP Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Sepsis: The puerperal / postpartum women who evolved with sepsis, needing support by invasive mechanical ventilation, were evaluated and monitored with Electrical Impedance Tomography for ventilatory therapy. In order to obtain the images and quantification of the regional ventilatory distribution, two strips with 16 electrodes were connected around the thorax to capture an imperceptible and harmless electric current to the patient, generating, according to the pulmonary dynamics, an impedance power of variation. A flow sensor was positioned between the endotracheal tube and the "Y" of the ventilator circuit and was responsible for capturing information about ventilatory mechanics. Data were sent simultaneously to a system (computer) with specific softwear in order to measure and quantify the regional distribution of pulmonary ventilation and perfusion, as well as their correlation.
  Interventions: Other: Sepsis
- HELLP Syndrome: The puerperal / postpartum women who evolved with HELLP syndrome, needing support by invasive mechanical ventilation, were evaluated and monitored with Electrical Impedance Tomography for ventilatory therapy. In order to obtain the images and quantification of the regional ventilatory distribution, two strips with 16 electrodes were connected around the thorax to capture an imperceptible and harmless electric current to the patient, generating, according to the pulmonary dynamics, an impedance power of variation. A flow sensor was positioned between the endotracheal tube and the "Y" of the ventilator circuit and was responsible for capturing information about ventilatory mechanics. Data were sent simultaneously to a system (computer) with specific softwear in order to measure and quantify the regional distribution of pulmonary ventilation and perfusion, as well as their correlation.
  Interventions: Other: HELLP Syndrome
- Respiratory Distress Syndrome, Adult: The puerperal / postpartum women who evolved with Adult Respiratory Distress Syndrome, needing support by invasive mechanical ventilation, were evaluated and monitored with Electrical Impedance Tomography for ventilatory therapy. In order to obtain the images and quantification of the regional ventilatory distribution, two strips with 16 electrodes were connected around the thorax to capture an imperceptible and harmless electric current to the patient, generating, according to the pulmonary dynamics, an impedance power of variation. A flow sensor was positioned between the endotracheal tube and the "Y" of the ventilator circuit and was responsible for capturing information about ventilatory mechanics. Data were sent simultaneously to a system (computer) with specific softwear in order to measure and quantify the regional distribution of pulmonary ventilation and perfusion, as well as their correlation.
  Interventions: Other: Respiratory Distress Syndrome Adult

INTERVENTIONS:
Other: Sepsis — Evaluation and monitoring with Electrical Impedance Tomography in order to conduct ventilatory therapy.
  Groups: Sepsis
Other: HELLP Syndrome — Evaluation and monitoring with Electrical Impedance Tomography in order to conduct ventilatory therapy.
  Groups: HELLP Syndrome
Other: Respiratory Distress Syndrome Adult — Evaluation and monitoring with Electrical Impedance Tomography in order to conduct ventilatory therapy.
  Groups: Respiratory Distress Syndrome, Adult

SUMMARY:
Introduction: Electrical Impedance Tomography (TIE) consists of an equipment that enables the visualization / quantification in real time of the regional distribution of ventilation and pulmonary perfusion, as well as of ventilatory mechanics. Used on the edge of the bed, it is easy to move, non-invasive, allowing a momentary or continuous assessment, guiding the conduct in a safe and precise way through the electrical impedance technology. It is important to note that, in addition to ensuring the efficacy of the patient's behavior, the TIE supports the most diverse types of studies to be performed. These include those based on the effectiveness of the use of the method in the most diverse pulmonary dysfunctions, in the adjustment of the mechanical ventilation and in the average time of hospitalization. Objective: To evaluate the pulmonary function of patients in invasive mechanical ventilation through SIT. Method: This research was carried out in compliance with the National Health Council's Guidelines for Research Involving Human Beings (466/12). The study was a prospective longitudinal clinical-experimental type in which all patients (occasional sampling) used mechanical ventilation and were hospitalized in the Adult Intensive Care Unit (ICU) of the Santa Casa de Misericórdia Foundation of Pará, and they developed sepsis with pulmonary repercussions; (DEHG) / HELLP Syndrome and Adult Respiratory Distress Syndrome (ARDS) and who met the inclusion criteria were evaluated and monitored with TIE to perform ventilatory therapy according to the research objectives. The research was carried out in the city of Belém, in the state of Pará, in the adult ICU of the FSCMP. As inclusion criterion, the patient should be in the FSCMP adult Intensive Care Unit (ICU), under mechanical invasive ventilation, previously authorized by the family through the Informed Consent Form to participate in the study.

DETAILED DESCRIPTION:
A prospective longitudinal clinical-experimental study was carried out in which 30 postpartum / postpartum women who developed complications of their clinical condition, needing support by invasive mechanical ventilation, development of sepsis with pulmonary repercussion, Specific Pregnancy Disease ( SDP), HELLP syndrome or ARDS were evaluated and monitored with Electrical Impedance Tomography for conduction of ventilatory therapy. In order to obtain the images and quantification of the regional ventilatory distribution, two tapes with 16 electrodes were connected by means of an adhesive tape, one for each band, around the thorax and aligned in a plane corresponding to a cross section with emission of an electric current imperceptible and harmless to the patient, generating, according to the pulmonary dynamics, a variation of electrical impedance, consequently a gradient of electrical resistivity. A flow sensor positioned between the endotracheal tube and the "Y" of the ventilator circuit, responsible for capturing ventilatory mechanic information, and a reference cable positioned by an electrocardiographic monitoring electrode, in the abdominal region or in the region from the shoulders. The data were sent simultaneously to a system (computer) with specific softwear in order to measure and quantify the regional distribution of pulmonary ventilation and perfusion, as well as its correlation in patients under mechanical ventilation. All experimental values were presented as mean ± standard deviation (SD). The study was of the experimental type, and the descriptive statistic was used to characterize the sample. Statistical analysis was performed with GraphPad Prism 5.0. The P value <0.05 was considered statistically significant. The results were placed in spreadsheets and graphs created with GraphPad Prism 5.0 (GraphPad Software, San Diego, California, USA).

ELIGIBILITY:
Inclusion Criteria: the patient should:

* To be admitted to the Adult Intensive Care Unit (ICU) of the FSCMP;
* Being in the postpartum/puerperium period;
* To evolve with complications of its clinical condition: sepsis with pulmonary repercussions, Specific Disease of Pregnancy (SDP), HELLP syndrome or ARDS;
* Support by invasive mechanical ventilation;
* To be previously authorized by the family to participate in the study through the WICF.

Exclusion Criteria:

* Being a cardiac pacemaker;
* Pregnant women in any period of gestation who develop complications of their clinical condition and need support through invasive ventilation.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postpartum women without age limits
Study Population: The sample of this research will be constituted by puerperas hospitalized in the adult ICU of the FSCMP from September 2017 to May 2018, and evolved with the diagnosis of ARDS, HELLP syndrome or sepsis, being sedated and requiring invasive mechanical ventilation in the assisted mode -controlled during his period of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Correlation of the driving pressure with the survival of puerperae under mechanical ventilation by electrical impedance tomography | Data will be collected 3 times a day in the morning, evening and evening hours until the conclusion of the study, with a mean of 3 to 5 days of monitoring by electrical impedance tomography
  For the delimitation of the information collection of postpartum women submitted to invasive mechanical ventilation for having evolved with HELLP syndrome, sepsis or respiratory distress syndrome, and ventilatory data were collected from the data sheet of the Electrical Impedance Tomography, containing data from the regional distribution of (Cst) of the respiratory system, final expiratory positive pressure (PEEP) and Platelet Pressure (Pplatô), as well as ventilatory parameters data: Ventilatory mode and mode, PEEP, VT, Inspiratory Time (I), Inspired Fraction of Oxygen (FiO2), Sensitivity (Sens.), Of hospitalized patients in the period of collections. After a retrospective survey of the sample, data were collected from patients who were in the Intensive Care Unit, while they were on invasive mechanical ventilation and monitored by Electrical Impedance Tomography.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Brenner DJ. Radiation risks potentially associated with low-dose CT screening of adult smokers for lung cancer. Radiology. 2004 May;231(2):440-5. doi: 10.1148/radiol.2312030880. PMID 15128988
- [Result] Cinnella G, Grasso S, Raimondo P, D'Antini D, Mirabella L, Rauseo M, Dambrosio M. Physiological Effects of the Open Lung Approach in Patients with Early, Mild, Diffuse Acute Respiratory Distress Syndrome: An Electrical Impedance Tomography Study. Anesthesiology. 2015 Nov;123(5):1113-21. doi: 10.1097/ALN.0000000000000862. PMID 26397017
- [Result] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Result] Frerichs I, Hinz J, Herrmann P, Weisser G, Hahn G, Dudykevych T, Quintel M, Hellige G. Detection of local lung air content by electrical impedance tomography compared with electron beam CT. J Appl Physiol (1985). 2002 Aug;93(2):660-6. doi: 10.1152/japplphysiol.00081.2002. PMID 12133877
- [Result] Frerichs I, Dargaville PA, Dudykevych T, Rimensberger PC. Electrical impedance tomography: a method for monitoring regional lung aeration and tidal volume distribution? Intensive Care Med. 2003 Dec;29(12):2312-2316. doi: 10.1007/s00134-003-2029-z. Epub 2003 Oct 18. PMID 14566457
- [Result] Jubran A. Advances in respiratory monitoring during mechanical ventilation. Chest. 1999 Nov;116(5):1416-25. doi: 10.1378/chest.116.5.1416. PMID 10559107
- [Result] Matthay MA, Zemans RL. The acute respiratory distress syndrome: pathogenesis and treatment. Annu Rev Pathol. 2011;6:147-63. doi: 10.1146/annurev-pathol-011110-130158. PMID 20936936
- [Result] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Result] Pearce MS, Salotti JA, Little MP, McHugh K, Lee C, Kim KP, Howe NL, Ronckers CM, Rajaraman P, Sir Craft AW, Parker L, Berrington de Gonzalez A. Radiation exposure from CT scans in childhood and subsequent risk of leukaemia and brain tumours: a retrospective cohort study. Lancet. 2012 Aug 4;380(9840):499-505. doi: 10.1016/S0140-6736(12)60815-0. Epub 2012 Jun 7. PMID 22681860
- [Result] Pesenti A, Musch G, Lichtenstein D, Mojoli F, Amato MBP, Cinnella G, Gattinoni L, Quintel M. Imaging in acute respiratory distress syndrome. Intensive Care Med. 2016 May;42(5):686-698. doi: 10.1007/s00134-016-4328-1. Epub 2016 Mar 31. PMID 27033882
- [Result] Reinius H, Borges JB, Freden F, Jideus L, Camargo ED, Amato MB, Hedenstierna G, Larsson A, Lennmyr F. Real-time ventilation and perfusion distributions by electrical impedance tomography during one-lung ventilation with capnothorax. Acta Anaesthesiol Scand. 2015 Mar;59(3):354-68. doi: 10.1111/aas.12455. Epub 2015 Jan 5. PMID 25556329